CLINICAL TRIAL: NCT05133193
Title: Efficacy and Safety of 14-day Concomitant Therapy for Refractory Helicobacter Pylori Infection：A Pilot Study
Brief Title: Efficacy and Safety of 14-day Concomitant Therapy for Refractory Helicobacter Pylori Infection
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shandong University (Other)
Responsible Party: Principal Investigator, Xiuli Zuo, Director of Qilu Hospital gastroenterology department, Shandong University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020-SDU-QILU-G057
Record Dates: First submitted 2021-11-13; First posted 2021-11-24 (Actual); Last update posted 2021-11-26 (Actual); Status verified 2021-11

CONDITIONS: Helicobacter Pylori Infection
Keywords: Concomitant Therapy,Rescue treatment
MeSH Terms: interventions — Anti-Bacterial Agents

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 14d concomitant therapy (Experimental): The eligible patients received 14-day concomitant therapy, including vonoprazan and three kinds of antibiotics according to the previous eradication regimens and antibiotic use. Antibiotics are selected from Amoxicillin, Tetracycline, Furazolidone, Levofloxacin, Clarithromycin, Tinidazole, Metronidazole.
  Interventions: Drug: three kinds of antibiotics

INTERVENTIONS:
Drug: three kinds of antibiotics — All patients were educated carefully about the medical instructions, including the duration of treatment, possible side effect, the necessity of completing the full 14-day course.
  Other Names: antibiotics

SUMMARY:
The purpose of this study is to evaluate efficacy of a 14-day concomitant therapy for the third-line treatment of Helicobacter pylori infection, and whether it is safe while maintaining an ideal eradication rates.

DETAILED DESCRIPTION:
Helicobacter pylori infects half of the world's population. H.pylori eradication is an effective approach to reduce the risk of developing gastric cancer. However, eradication rates of first-line therapy decreased over years due to the rapidly increasing antibiotic resistance of H. pylori worldwide. An ideal rescue therapeutic regimen to cure refractory H.pylori infection is currently warranted.

Few published paper evaluated the efficacy of 14-day furazolidone containing concomitant therapy in the third line treatment. This study aims to propose a new concomitant therapy for the patients with three or more treatment failure, and then evaluates whether adverse effects are tolerable. .

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-70 years were recruited for this study if they had failed at least three rounds of anti- H. pylori therapies.

Exclusion Criteria:

* Patients treated with H2-receptor antagonist, PPI, vonoprazan, bismuth and antibiotics in the previous 4 weeks
* Patients with gastorectomy, acute GI bleeding and advanced gastric cancer,
* History of allergy to any of the drugs used in the study,
* Severe concomitant cardiovascular, respiratory, or endocrine diseases, clinically significant renal or hepatic disease, hematologic disorders and any other clinically significant medical condition that could increase risk,
* Currently pregnant or lactating,
* Severe neurologic or psychiatric disorders,
* Alcohol abuse or drug addiction,
* Patients with compliance lower than 90% in any previous treatment,
* Inability to provide informed consent and other situations that could interfere with the examination or therapeutic protocol.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-11-20 (Estimated); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
Eradication rate | 6 month
  Six weeks after completion of treatment,number of patients get H.pylori eradicated will be investigated.Then eradication rate will be calculated by using intention-to-treat analysis and per-protocol analysis

SECONDARY OUTCOMES:
The rates of adverse events | 6 month
  At the follow-up,adverse events complained by patients will be recorded by an inde pendent researcher, meanwhile a 8point visual analog scale (VAS) was used to evaluate severity of adverse events.
Compliance | 6 month
  Compliance was evaluated by assessing the total pills patients have taken.Compliance was defined as good when more than 80% or less than 120% of the total pills were taken.